CLINICAL TRIAL: NCT00494806
Title: The Effects of Rocking Chair Motion on Postoperative Ileus Duration, Subjective Pain and Time to Discharge Following Abdominal Surgery
Brief Title: Effects of Rocking on Postoperative Ileus Duration Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2004-0887
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-07

CONDITIONS: Abdominal Cancer
Keywords: Postoperative Ileus (POI); Rocking Chair; Abdominal Cancer

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rocking Group (Experimental): Patients rocked in a rocking chair in 10-20 minute increments for at least one hour per day beginning on the first day after surgery. Activity was increased each day and continued until passage of first postoperative flatus.
  Interventions: Other: Rocking Chair Intervention
- Standard Care (No Intervention): Standard care group got out of bed and sat in a non-rocking chair and ambulated beginning the first day after surgery. Activity was increased each day and continued until passage of first postoperative flatus.

INTERVENTIONS:
Other: Rocking Chair Intervention — Patient out of bed rocking in a rocking chair at a constant rate of one rock cycle per second (back and forth), in ten to twenty minute increments, for at least sixty minutes per day or 3600 rock cycles and ambulate at least twice per day beginning the first postoperative day.
  Arms: Rocking Group

SUMMARY:
Primary Objective:

1. Compare the duration of postoperative ileus (POI) duration (time to first flatus), subjective reports of surgical and gas pain, postoperative pain medication (total milligrams per 24 hours) and postoperative recovery time(length of stay) between two groups of abdominal surgery cancer patients receiving either standard postoperative care or standard care plus the rocking intervention.

DETAILED DESCRIPTION:
Ileus is a lack of bowel function that can cause colic, vomiting, and/or constipation. Research has shown that bowel function slows down and possibly stops working for a short period of time after surgery, usually for 5-7 days. Patients report pain and discomfort from the gas that builds up in their bowel until the time the bowel begins working properly after surgery. During the period the bowel is not working after surgery, patients cannot leave the hospital until their physician is sure that their bowel function has returned. The return in bowel function is usually signaled by the passage of gas from the rectum.

The main method used to help the return of bowel function is to have patients get out of bed, sit in a chair, and begin walking the first day after surgery and increase the time sitting in the chair and walking every day. However, it is not clear that the sitting in a chair and walking are the best methods to assist in a faster return of bowel function.

One method that shows promise in helping the return of bowel function after abdominal surgery is rocking in a rocking chair. Rocking chair motion has demonstrated an earlier return of normal bowel function in mothers after C-Section and women after abdominal hysterectomy (Moore et al.,1995; Thomas et al., 1990). Rocking also has been used to decrease pain, the amount of pain medication needed, and the time spent in the hospital after abdominal surgery.

If you agree to take part in this study, you will be randomly assigned to one of two groups (Group A or B). Participants in Group A will use the rocking chair method. Participants in Group B will not use the rocking chair method. There is an equal chance of being assigned to either group.

Before you take part in this study, you will be asked to complete a survey about the amount of pain you are currently experiencing (the Brief Pain Inventory-Short Form). It should take about 10 minutes to complete the Brief Pain Inventory-Short Form. Completing the pain inventory before your surgery will allow for a better comparison of your pre and postoperative surgical and gas pain. You will be asked to provide some information such as your age and marital status that will be recorded on a coded data sheet. You will also receive an instruction sheet that describes what you need to do in order to participate in the study (Instruction to Subjects Sheet). The study investigator will also demonstrate to those chosen for the rocking group the correct method to rock in the rocking chair and allow them time to practice. He will also demonstrate the correct way to wear the gait belt with the pedometer attached to it.

Participants in Group A will get out of bed beginning the first day after surgery, sit in a rocking chair (at least twice per day), and rock backward and forward at a constant rate of 1 backward and forward rock per second in 10-20 minute increments. This will be done for at least 60 minutes (1 hour) per day. Participants in Group A will also be asked to begin walking at least twice per day beginning the first day after surgery.

Participants in Group B will get out of bed beginning the first day after surgery and sit in a non rocking chair (at least twice per day) for at least sixty minutes. Group B will also be asked to begin walking at least twice per day.

Both groups will wear a pedometer attached to a gait belt worn around their waist in order to record the number of steps taken in a 24-hour period of time. A pedometer will also be attached to each rocking chair in order to record the number of rocks in a 24-hour period. Participants in each group will be encouraged by the research staff to increase the time spent rocking, sitting in the non-rocking chair, and walking each day. You will be given pain medication as needed.

All participants will be given a pencil and pad to note the date and time that they first pass gas from their rectum. A calendar and clock is available in all patient rooms. Every morning, the study investigator will visit you and ask if you have passed gas, record the number of rocks and steps recorded by the pedometers, reset the pedometers, have you complete a Brief Pain Inventory-Short Form pain evaluation, and check on the total amount of pain medication you have received over the last 24 hours. You may increase the time spent rocking and walking as you desire and are encouraged to do so.

If for any reason, you cannot tolerate rocking in a rocking chair, sitting in a non rocking chair or walking because of discomfort or any other reason, you will be removed from the study without penalty.

There is no follow-up testing for this study. The length of this study is from the first day after your surgery until you actually pass gas from the rectum. This time could range from 5 to 7 days after your operation.

This is an investigational study. There are no drugs involved with this study. Rocking, non rocking chairs, and gait belts will be provided by M. D. Anderson and the pedometers by the study investigator at no charge to the participants during the study. A total of 66 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Post abdominal surgical cancer patient, undergoing abdominal surgery
2. Over 21 years of age.
3. Ambulatory.
4. Cognitively intact.
5. Scheduled to have epidural analgesia with fentanyl or dilaudid and/or patient controlled analgesia with morphine or dilaudid as their primary mode of postoperative pain control.

Exclusion Criteria:

1. Postoperative abdominal surgical cancer patient less than 21 years of age.
2. Are not ambulatory.
3. Are not cognitively intact.
4. Have any of the following: severe neuromuscular disease, cardiovascular disease, pacemakers, inner-ear disturbances, known peripheral vascular disease that interferes with ambulation, are on sympathetic inhibitory or mood altering drugs. All patients will have epidural and/or patient controlled analgesia as their primary mode of postoperative pain control and those who do not will be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2005-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Massey, RN, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 11/18/05 through 03/05/07. All participants recruited at UT MD Anderson Cancer Center, prior to surgery during their preoperative evaluation in the Anesthesia Assessment and Preoperative centers.
Pre-assignment Details: There were no enrolled participates excluded from the trial prior to assignment to groups. All patients approached accepted participation into the study.
Groups:
- Rocking Chair: Patients rocked in a rocking chair in 10-20 minute increments for at least one hour per day beginning on the first day after surgery. Activity was increased each day and continued until passage of first postoperative flatus.
Period: Overall Study
Arm/Group | Rocking Chair | Standard Care
Started | 34 | 32
Completed | 34 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rocking Chair | Standard Care | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 31 | 64
  >=65 years | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 56.2 (10.1) | 54.8 (11.4) | 55.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 13 | 33
  Male | 14 | 19 | 33
Region of Enrollment [Number; unit: participants]
  United States | 34 | 32 | 66

OUTCOME MEASURES:

1. Primary Outcome: Time to First Postoperative Flatus in Days Was the End of Postoperative Ileus (POI) Indicator.
Description: Time from end of surgical procedure until passage of first postoperative flatus was used as an indicator for resolution of postoperatve ileus (POI).
Time Frame: Daily from first day after surgical procedure to passage of first flatus (up to 5 - 7 days post surgery).
Population: Intention to treat (ITT) method was used.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Rocking Chair | Standard Care
Number analyzed (Participants) | 34 | 32
Days | 3.16 (0.86) | 3.88 (0.80)
Statistical Analysis 1: Comparison: Rocking Chair vs Standard Care; No differences in time to first flatus between the rocking and non rocking groups is the null hypothesis. Sample size calculations by setting the criterion for significance at .05, two-tailed test (an effect in either directions was accepted), and power at .80. A total sample of 54 participants was determined necessary to yield statistically significant results (27 in Group A and 27 in Group B); Test type: Superiority or Other; p < 0.05, t-test, 2 sided; df = 64; Mean Difference (Final Values) = 0.7279, 95% CI [0.3174 to 1.1383], Standard Error of Mean .15 — Relative risk not calculated

ADVERSE EVENTS:
Arm/Group | Rocking Chair | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32
Other Adverse Events (participants affected / at risk) | 0/34 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No